CLINICAL TRIAL: NCT04665154
Title: A First-in-human, Randomized, Subject-blinded, Placebo-controlled, Single Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of MAS825 in Healthy Volunteers
Brief Title: A First-in-human Study to Investigate the Safety, Tolerability and Pharmacokinetics of MAS825 in Healthy Volunteers
Acronym: MAS-FIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMAS825A02101
Record Dates: First submitted 2020-11-30; First posted 2020-12-11 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MAS825 dose A (Experimental): single i.v. dose
  Interventions: Drug: MAS825
- MAS825 dose B (Experimental): single s.c. dose
  Interventions: Drug: MAS825
- Placebo dose A (Placebo Comparator): single i.v. dose
  Interventions: Drug: Placebo
- Placebo dose B (Placebo Comparator): single s.c. dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MAS825 — single dose i.v. and s.c.
  Arms: MAS825 dose A; MAS825 dose B
Drug: Placebo — single dose i.v. and s.c.
  Arms: Placebo dose A; Placebo dose B

SUMMARY:
The study is conducted to investigate the safety, tolerability and pharmacokinetics of MAS825 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

• Healthy male and female subjects 18 to 45 years of age included, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant
* A history of ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold test
* Fasting LDL > 160 mg/dL, at screening.
* Subjects in cohorts D1 and D2 (Japanese cohorts) must be of first to third generation Japanese ethnic origin.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | up to day 253
  To assess the safety and tolerability of single i.v./s.c. doses of MAS825

SECONDARY OUTCOMES:
Concentrations of anti-MAS825 antibodies | up to day 197
  To assess immunogenicity (IG) of MAS825
Pharmacokinetic parameters of MAS825: Maximum Plasma Concentration [Cmax] | up to day 197
  Cmax is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass x volume-1)
Pharmacokinetic parameters of MAS825: Time to reach maximum concentration [Tmax] | up to day 197
  Tmax is the time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration (time)
Pharmacokinetic parameters of MAS825: AUClast | up to day 197
  The AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1)
Pharmacokinetic parameters of MAS825: AUCinf | up to day 197
  The AUC from time zero to infinity (mass x time x volume-1)
Pharmacokinetic parameters of MAS825: T1/2 | up to day 197
  The elimination half-life associated with the terminal slope (lambda_z) of a semi logarithmic concentration-time curve (time). Use qualifier for other half-lives
Pharmacokinetic parameters of MAS825: CL | up to day 197
  CL is the systemic (or total body) clearance from plasma (or serum or blood) following intravenous administration [volume / time]
Pharmacokinetic parameters of MAS825: Vz | up to day 197
  Vz is the volume of distribution during the terminal elimination phase following intravenous administration [volume]
Pharmacokinetic parameters of MAS825: Vz/F | up to day 197
  Vz/F is the apparent volume of distribution during the terminal elimination phase following s.c. administration (associated with λz) (volume)
Pharmacokinetic parameters of MAS825: Vss | up to day 197
  Vss is the volume of distribution at steady state following intravenous administration [volume]
Pharmacokinetic parameters of MAS825: CL/F | up to day 197
  CL/F is the apparent systemic (or total body) clearance from plasma (or serum or blood) following s.c. administration [volume / time]

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Novartis Investigative Site, Tempe, Arizona
  - Novartis Investigative Site, Overland Park, Kansas
- Novartis Investigative Site, Mere Way, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com